CLINICAL TRIAL: NCT00238355
Title: Phase II Trial of Voriconazole Plus Caspofungin for the Initial Treatment of Invasive Fungal Infections
Brief Title: Voriconazole and Caspofungin Acetate in Treating Invasive Fungal Infections in Patients With Weakened Immune Systems
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: competing study at site
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000445848; OHSU-HEM-0346-L (Other: OHSU Knight Cancer Institute); OHSU-IRB-1379 (Other: OHSU IRB)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Infection; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: infection; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Infections | interventions — Caspofungin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Voriconazole plus Caspofungin (Experimental)
  Interventions: Drug: caspofungin acetate; Drug: voriconazole

INTERVENTIONS:
Drug: caspofungin acetate — 70 mg iv x 1 on day 1 (loading dose), followed by 50 mg iv daily on day 2 through day 84.
Drug: voriconazole — 6mg/kg iv q12 hours x 2 doses OR 400mg po q12hours on day 1 (loading doses. Maintenance doses on day 2 through day 84 may be either 4 mg/kg iv q12 hours, or 200 mg po q12 hours (at least one hour before or after meals).

SUMMARY:
RATIONALE: Voriconazole and caspofungin acetate may control invasive fungal infections in patients who have weakened immune systems.

PURPOSE: This phase II trial is studying how well giving voriconazole together with caspofungin acetate works in treating invasive fungal infections in patients with weakened immune systems.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 12-week complete and partial response rate in immunocompromised patients with invasive fungal infections treated with voriconazole and caspofungin acetate.

Secondary

* Determine the 12-week survival rate in patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: Patients receive voriconazole orally or IV over 1 hour twice daily and caspofungin acetate IV over 1 hour once daily on days 1-84. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of probable or definite invasive fungal infection with 1 of the following organisms:

  * Aspergillus species
  * Fusarium species
  * Scedosporium species (Pseudallescheria boydii)
  * Other dematiaceous molds
* The following diagnosis are not allowed:

  * Zygomycetes (Mucor or Rhizopus species)
  * Chronic aspergillosis
  * Aspergilloma
  * Allergic bronchopulmonary aspergillosis
* Must be immunocompromised

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* At least 72 hours

Hematopoietic

* Not specified

Hepatic

* AST < 5 times upper limit of normal (ULN)
* Bilirubin < 5 times ULN
* Alkaline phosphatase < 5 times ULN
* No Child-Pugh class C cirrhosis

Renal

* Creatinine clearance ≥ 50 mL/min

Pulmonary

* No mechanical ventilation

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No hypersensitivity to azoles, caspofungin acetate, or their components
* No history of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 14 days since prior therapeutic antifungal therapy of ≥ 1 week duration
* More than 14 days since prior and no concurrent administration of any of the following medications:

  * Terfenadine
  * Astemizole
  * Cisapride
  * Pimozide
  * Quinidine
  * Sirolimus
  * Rifampin
  * Carbamazepine
  * Long-acting barbiturates
  * Rifabutin
  * Ergot alkaloids (i.e., ergotamine and dihydroergotamine)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Strasfeld, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole Plus Caspofungin: Voriconazole: 6mg/kg iv q12 hours x 2 doses OR 400mg po q12hours on day 1 (loading doses). Maintenance doses on day 2 through day 84 may be either 4 mg/kg iv q12 hours, or 200 mg po q12 hours
  Caspofungin: 70 mg iv x 1 on day 1 (loading dose), followed by 50 mg iv daily on day 2 through day 84.
Period: Overall Study
Arm/Group | Voriconazole Plus Caspofungin
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole Plus Caspofungin
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.916 (15.370)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete or Partial Response Rate to the Combination of Voriconazole and Caspofungin at 12 Weeks.
Description: Patients will be followed through day 84 (12 weeks), regardless of continuation of study drugs. Complete response: Resolution of all clinical signs and symptoms and more than 90 percent of the lesions due to invasive fungus that were visible by radiology. Partial response: Clinical improvement and greater than 50 percent improvement in the lesions due to invasive fungus that were visible by radiology.
Time Frame: 12 weeks after starting treatment
Measure: Number; unit: Participants
Arm/Group | Voriconazole Plus Caspofungin
Number analyzed (Participants) | 13
Participants | 4

2. Secondary Outcome: Survival at 12 Weeks
Description: Defined as the number of evaluable subjects alive at 12 weeks (84 days) following registration.
Time Frame: up to 12 weeks
Population: 3 subjects were not evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Voriconazole Plus Caspofungin
Number analyzed (Participants) | 10
participants | 4

ADVERSE EVENTS:
Arm/Group | Voriconazole Plus Caspofungin
Serious Adverse Events (participants affected / at risk) | 10/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole Plus Caspofungin (N=13)
Sepsis (Blood and lymphatic system disorders) | 1
Liver and Renal failure (Renal and urinary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Abdominal Pain (General disorders) | 2
Altered Mental State (Psychiatric disorders) | 1
Cerebral Hemorrhage (Vascular disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Disease Progression (General disorders) | 2
Intracerebral Hemorrhage (Vascular disorders) | 1
Pulmonary Infection (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No